CLINICAL TRIAL: NCT05396313
Title: Development and Validation of Predictive Models for Mortality After CIED Implantation
Brief Title: Prediction of Mortality After CIED Implantation (PM-CIED)
Acronym: PM-CIED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Yixiu Liang, Doctor, Shanghai Zhongshan Hospital
Other Study IDs: PM-CIED
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Heart Failure, Systolic; Sudden Cardiac Death
MeSH Terms: conditions — Heart Failure, Systolic; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Zhongshan Hospital cohort: Patients receiving CIED implantation at Zhongshan Hospital
  Interventions: Device: CRT/ICD
- Fuwai Hospital cohort: Patients receiving CIED implantation at Fuwai Hospital
  Interventions: Device: CRT/ICD
- Shanghai Chest Hospital cohort: Patients receiving CIED implantation at Shanghai Chest Hospital
  Interventions: Device: CRT/ICD

INTERVENTIONS:
Device: CRT/ICD — The patients received implantation of CRT/ICD.

SUMMARY:
The study aims to develop and validate predictive models for the mortality of patients receiving CIED (including CRT and ICD) implantation.

DETAILED DESCRIPTION:
The study aims to develop and validate predictive models for the mortality of patients receiving cardiovascular implantable electronic devices (CIED) [including cardiac resynchronization therapy (CRT) and implantable cardioverter defibrillator (ICD)] implantation, with traditional statistical analysis and machine learning algorithms.

ELIGIBILITY:
Inclusion Criteria:

* all patients who received implantation of CRT/ICD

Exclusion Criteria:

* patients who received generator placement of CRT/ICD

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients who received CRT/ICD implantation for heart failure or high risk of sudden cardiac death (SCD).
Sampling Method: Non-Probability Sample
Enrollment: 1618 (Estimated)
Dates: Start 2004-08 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 3 years
  All-cause death

CONTACTS AND LOCATIONS:
Overall Officials: Yixiu Liang, MD, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pan L, Liu X, Zhu L, Yu Z, Wang J, Li X, Zhang W, Li R, Wang Z, Lu H, Yang S, Li P, Su Y, Hua W, Liang Y. Machine Learning-Based Prognostic Models for Mortality in Patients Receiving Implantable Cardioverter Defibrillators. Pacing Clin Electrophysiol. 2025 Aug;48(8):906-916. doi: 10.1111/pace.70008. Epub 2025 Jul 8. PMID 40625105